CLINICAL TRIAL: NCT03630341
Title: Adding L-Carnitine to Clomiphene Citrate for Induction of Ovulation in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCCC
Record Dates: First submitted 2018-08-04; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): This group will receive oral clomiphene citrate 50 mg tablet, two times per day from the third day of the cycle until the seventh day of the cycle plus oral carnitine 1g tablet, three times per day from the third day until the day of the pregnancy test.
  Interventions: Drug: Clomiphene Citrate 50mg; Drug: L-carnitine
- control group (Active Comparator): This group will receive oral clomiphene citrate 50 mg tablet, two times per day from the third day of the cycle until the seventh day of the cycle plus oral placebo tablet, three times per day from the third day until the day of the pregnancy test.
  Interventions: Drug: Clomiphene Citrate 50mg; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Clomiphene Citrate 50mg — oral 50 mg tablets
Drug: L-carnitine — 1000 mg oral tablet
  Arms: study group
Drug: Placebo Oral Tablet — oral tablets identical to L-carnitine
  Arms: control group

SUMMARY:
Polycystic ovary syndrome is one of the most common endocrine disorders, affecting about 6-10% of women in their reproductive age. Anovulation and hyperandrogenism are often present together with hyperinsulinaemia and insulin resistance

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary infertility.
* Normal Hysterosalpingo-graphy
* Normal Semen analysis of the husband.

Exclusion Criteria:

* Patient's refusal.
* Male factors of infertility and/or abnormal Hysterosalpingo-graphy
* Hyperprolactinemia (prolactin ≥ 22 ng/dl).
* FSH on day 3 > 15 mIU/mL.
* Gross ovarian pathology diagnosed by ultrasound.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 1 month
  visible intra-uterine gestational sac, with a positive fetal heart beat, viewed during a transvaginal ultrasound (when the b-hCG concentration was more than 1500 IU/l)

IPD SHARING:
Plan to Share IPD: No